CLINICAL TRIAL: NCT04631029
Title: A Phase 1 Study of Entinostat in Combination With Atezolizumab / Carboplatin / Etoposide in Previously Untreated Extensive-Stage Small Cell Lung Cancer
Brief Title: Testing the Addition of an Anti-cancer Drug, Entinostat, to the Usual Chemotherapy and Immunotherapy Treatment (Atezolizumab, Carboplatin and Etoposide) for Previously Untreated Aggressive Lung Cancer That Has Spread
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-09916; NCI-2020-09916 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10399 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10399 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2020-11-14; First posted 2020-11-17 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma; Malignant Solid Neoplasm; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — atezolizumab; Carboplatin; entinostat; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (carboplatin, etoposide, atezolizumab, entinostat) (Experimental): INDUCTION THERAPY: Patients receive carboplatin IV over 30-60 minutes on day 1, etoposide IV over 60 minutes on days 1-3, atezolizumab IV over 30-60 minutes on day 1, and entinostat PO on days 1, 8, and 15. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive atezolizumab IV over 30 minutes on day 1 and entinostat PO on days 1, 8, and 15. Treatment repeats every 21 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Atezolizumab; Drug: Carboplatin; Drug: Entinostat; Drug: Etoposide

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS-275; SNDX-275
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP16

SUMMARY:
This phase I trial seeks to find out the best dose, possible benefits and/or side effects of entinostat in combination with atezolizumab, carboplatin and etoposide for the treatment of previously untreated aggressive lung cancer that has spread (extensive-stage small cell lung cancer). Entinostat and etoposide may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Carboplatin is a chemotherapy drug that attaches to deoxyribonucleic acid (DNA) and may kill tumor cells. Giving entinostat in combination with atezolizumab, carboplatin and etoposide may work better than atezolizumab, carboplatin and etoposide alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of entinostat in combination with carboplatin, etoposide, and atezolizumab.

II. To determine safety and tolerability of adding entinostat to carboplatin / etoposide / atezolizumab for extensive-stage small cell lung cancer (ES-SCLC).

III. To determine the feasibility of administering entinostat concomitantly with atezolizumab, carboplatin, and etoposide as determined by the proportion of patients who receive 3 or more cycles of the combination.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To determine the proportion of patients who are alive and without disease progression at 9 months (9 month progression free survival [PFS]) after starting entinostat, carboplatin, etoposide, and atezolizumab.

EXPLORATORY OBJECTIVES:

I. To estimate the clinical activity of entinostat plus carboplatin/etoposide/atezolizumab as determined by response rate (RR), progression free survival (PFS), and overall survival (OS).

II. To explore the prevalence of cyclic adenosine monophosphate (cAMP) response element binding protein (CREB) binding protein (CREBBP)/ histone acetyltransferase p300 (EP300) mutations in newly diagnosed ES-SCLC population.

III. To explore the relationship between CREBBP/EP300 mutations and clinical outcomes.

IV. To explore immune biomarkers that may predict response to atezolizumab and entinostat and changes in these biomarkers over the course of study treatment.

V. To explore entinostat exposure-response relationships with toxicity and clinical outcomes (PFS and OS).

VI. To evaluate baseline atezolizumab clearance as an early biomarker for OS and to assess the relationship between atezolizumab time-varying clearance, cachexia and clinical outcomes (PFS and OS).

OUTLINE: This is a dose-escalation study of entinostat.

INDUCTION THERAPY: Patients receive carboplatin intravenously (IV) over 30-60 minutes on day 1, etoposide IV over 60 minutes on days 1-3, atezolizumab IV over 30-60 minutes on day 1, and entinostat orally (PO) on days 1, 8, and 15. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive atezolizumab IV over 30 minutes on day 1 and entinostat PO on days 1, 8, and 15. Treatment repeats every 21 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 2 years, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed extensive stage SCLC (ES-SCLC) or other solid tumors for which carboplatin and etoposide are considered appropriate therapy
* No prior systemic therapy for extensive-stage, metastatic disease. Patients with prior limited stage disease who were treated with chemotherapy and concurrent radiation will be permitted to enroll as long as their previous treatment was 12 months or more prior to study enrollment
* Patients with treated brain metastases are eligible if they have stable symptoms and no ongoing requirement for corticosteroids as therapy for brain metastases
* Patients with untreated or progressive brain metastases (active brain metastases) are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy. There must be no ongoing requirement for corticosteroids as therapy for brain metastases
* Previous radiation, including whole brain radiation, is allowed >= 7 days of study registration. Stereotactic radiation therapy within 7 days is permitted
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. At least one measurable lesion should be extra-cranial and outside of any portal of irradiation
* Archival tissue must be available, or patients must be willing to undergo a new biopsy to provide pre-treatment tumor sample (no intervening chemotherapy treatment, tissue must be from current extensive-stage/metastatic diagnosis)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9.0 g/dL
* Platelets >= 100,000/mcL
* International normalized ratio (INR) < 1.5
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN). (This does not apply to patients with confirmed Gilbert's syndrome)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN, (if liver metastases present, can be up to 5 x ULN)
* Creatinine =< institutional ULN OR glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 (by the Cockcroft-Gault equation)
* Serum sodium >= 130 mmol/L
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* The effects of entinostat on the developing human fetus are unknown. For this reason and because histone deacetylase inhibitor (HDACi) agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, up to 5 months after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 5 months after completion of study treatment
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients with evidence of leptomeningeal metastases (either by imaging or central nervous system [CNS] fluid findings)
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to entinostat or other agents used in study
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because entinostat is HDACi agent with the potential for teratogenic or abortifacient effects and because of known teratogenic and abortifacient effects of cisplatin and etoposide. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with entinostat, and known risks with cisplatin and etoposide, breastfeeding should be discontinued if the mother is treated with entinostat. These potential risks may also apply to other agents used in this study
* Patients with a history of autoimmune disease (notable exceptions include hypothyroidism on thyroid replacement medication, type I diabetes, psoriasis or other cutaneous disease controlled with topical agents and without flare in 12 months requiring other treatment, celiac disease controlled with diet alone)
* Patients with a history of pulmonary fibrosis (history of radiation pneumonitis/fibrosis in the treatment field is permitted if stable and not requiring supplemental oxygen or corticosteroid use)
* Patients with prior history of allogeneic bone marrow or solid organ transplant
* Ongoing use of systemic corticosteroids or immunosuppressive agents within 14 days (inhaled corticosteroids, < 7 day course of prednisone for asthma/chronic obstructive pulmonary disease [COPD] exacerbation, or chronic low-dose supplemental steroids for adrenal insufficiency permitted)
* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents.

  * Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided the following requirements are met:

    * Minimum of 12 weeks from the first dose of anti-CTLA-4 and > 6 weeks from the last dose
    * No history of severe immune-related adverse effects from anti-CTLA-4 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] grade 3 and 4)
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2) within 6 weeks prior to study registration
* Patients taking bisphosphonate therapy for symptomatic hypercalcemia. Use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed
* Patients requiring treatment with a receptor activator of nuclear factor kappa-Β ligand (RANKL) inhibitor (e.g. denosumab) who cannot discontinue it before treatment with atezolizumab
* Patients requiring treatment with strong CYP3A inhibitors and inducers who cannot discontinue it before treatment with etoposide

  * Because the list of these agents are constantly changing, it is important to regularly consult a frequently updated list such as Facts and Comparisons or Lexicompt; medical reference texts such as the Physicians' Desk Reference may also provide this information
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* Patients with active tuberculosis (TB) are excluded
* Suspected or confirmed active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection (COVID-19).

  * Those with a history of COVID-19 are eligible if they meet all of the above eligibility criteria after clearance of COVID-19 by one of the following criteria:

    * 14 days have elapsed since symptom onset, the patient is afebrile, and symptoms are improving for at least 72 hours
    * Have 2 negative specimens collected at least 24 hours apart
* Severe infections within 2 weeks prior to study registration, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Received oral or intravenous (IV) antibiotics within 1 week prior to study registration. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 4 weeks prior to study registration or anticipation of need for a major surgical procedure during the course of the study. Common procedures such as biopsies, port insertions, and thoracenteses are allowed
* Administration of a live, attenuated vaccine within 4 weeks before study registration or anticipation that such a live, attenuated vaccine will be required during the study or up to 5 months after the last dose of atezolizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan D Gentzler, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Gentzler RD, Villaruz LC, Rhee JC, Horton B, Mock J, Hanley M, Kim K, Rudek MA, Phelps MA, Carducci MA, Piekarz R, Park KS, Bullock TN, Rudin CM. Phase I Study of Entinostat, Atezolizumab, Carboplatin, and Etoposide in Previously Untreated Extensive-Stage Small Cell Lung Cancer, ETCTN 10399. Oncologist. 2023 Nov 2;28(11):1007-e1107. doi: 10.1093/oncolo/oyad221. PMID 37555284

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: INDUCTION THERAPY: Patients receive carboplatin IV over 30-60 minutes on day 1, etoposide IV over 60 minutes on days 1-3, atezolizumab IV over 30-60 minutes on day 1, and entinostat 2 mg PO on days 1, 8, and 15. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive atezolizumab IV over 30 minutes on day 1 and entinostat PO on days 1, 8, and 15. Treatment repeats every 21 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dose Level 1
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dose Level 1
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 32 [18 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
Disease Stage [Count of Participants; unit: Participants] — Stage III disease is considered advanced disease. Stage IV disease is metastatic disease, which means the cancer has spread to other parts of the body. Participants with Metastatic (Stage IV) disease are considered to have worse disease than participants with Advanced (Sage III) disease.
  Participants
    Advanced (Stage III) disease | 1
    Metastatic (Stage IV) disease | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: The Bayesian optimal interval (BOIN) design will be used to find the MTD based on safety as determined by dose limiting toxicities.
Time Frame: Up to 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1
Number analyzed (Participants) | 3
Participants
  Completed Dose Level 1 without a dose-limiting toxicity | 1
  Experienced a dose limiting toxicity in Dose Level 1 | 2

2. Primary Outcome: Number of Participants Experiencing Grade 3 and 4 Adverse Events
Description: Defined by Common Terminology Criteria for Adverse Events version 5.0. Will be summarized by frequency and magnitude.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1
Number analyzed (Participants) | 3
Participants
  Grade 3 Adverse Events | 3
  Grade 4 Adverse Events | 2

3. Primary Outcome: Number of Participants Who Received 3 or More Cycles of the Combination of Entinostat, Atezolizumab, Carboplatin, and Etoposide
Description: The proportion of participants who received 3 or more cycles of the combination, will be calculated with a 90% confidence interval.
Time Frame: Up to cycle 4 (1 cycle = 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1
Number analyzed (Participants) | 3
Participants
  Received 3 or more cycles | 0
  Received 1 or 2 cycles | 3

4. Secondary Outcome: Progression Free Survival (PFS) Rate
Description: Defined as the proportion of patients alive and without disease progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Will be estimated with a 90% confidence interval. The Kaplan Meier estimator will be used to estimate survival curves.
Time Frame: Up to 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1
Number analyzed (Participants) | 3
Participants
  Alive without Disease Progression | 0
  Deceased by 2 months | 1
  Withdrew by 2 months | 2

ADVERSE EVENTS:
Time Frame: Up to 2 months
Arm/Group | Dose Level 1
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Lung infection (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Sepsis (Infections and infestations) | 1
Typhlitis (Gastrointestinal disorders) | 1
White blood cell count decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3)
Activated partial thromboplastin time prolonged (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 3
Atrial fibrillation (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatine kinase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Gastroesophageal reflux disease (GERD) (Gastrointestinal disorders) | 1
Hypertension (Vascular disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 2
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Platelet count decreased (Investigations) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
White blood cell decreased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT04631029/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT04631029/ICF_001.pdf